CLINICAL TRIAL: NCT00919334
Title: Control of Myopia Progression in Myopic Children Using Simultaneous Vision Approach
Brief Title: Myopia Control With Simultaneous Vision Approach
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Carly Lam, Head of School, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GRF5438/06M
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-07

CONDITIONS: Myopia
Keywords: Myopia progression; Myopia control; Simultaneous vision; Myopic defocus
MeSH Terms: conditions — Myopia | interventions — Lenses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- single vision soft contact lens (No Intervention): Single vision soft contact lenses with same materials of the DISC lens
- Defocus Incorporated Soft Contact (DISC) lens (Experimental): The use of DISC lens to slow down the progression of myopia
  Interventions: Device: Defocus Incorporated Soft Contact (DISC) lens

INTERVENTIONS:
Device: Defocus Incorporated Soft Contact (DISC) lens — Use of simultaneous vision bifocal soft contact lenses with myopic defocus to control the progression of myopia
  Other Names: myopia control; myopia progression; Simultaneous vision; bifocal contact lens
  Arms: Defocus Incorporated Soft Contact (DISC) lens

SUMMARY:
To determine if the 'Defocus Incorporated Soft Contact' (DISC) lens slows myopia progression in Hong Kong schoolchildren using simultaneous vision approach.

DETAILED DESCRIPTION:
The investigators hypothesize that the natural process of emmetropization in human is regulated by the equilibrium between the opposite hyperopic and myopic defocus. A sharp focus of retinal image (foveal fixation) is fundamental for co-ordination of the equilibrium. The DISC lens is a custom-made multi-zone bifocal soft contact lens which is based on simultaneously provides clear vision and defocus at all viewing distances. It comprises of correcting zones for correcting distant prescription(correction of refractive error, and defocusing zones to incorporate constant myopic defocus for slowing down myopia progression.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-13 years
* Myopia (SE) between -1D to -5D
* Astigmatism less than or equal to -1D
* Anisometropia: less than or equal to 1.25D
* aided VA (monocular): 0.00 log MAR or better
* willingness to wear contact lens constantly
* availability for follow-up for at least 2.5 years
* parents' understanding and acceptance
* willing to provide refractive status of grandparents

Exclusion Criteria:

* Severe ocular or systemic allergies
* Taking any medication that might have an impact on contact lens wear or that might influence the outcome of the clinical trial
* Ocular or systemic condition that might affect refractive development
* Strabismus at distance or near
* Prior use of bifocal or progressive lenses
* Prior use of rigid gas permeable lenses and Ortho-K lenses

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2007-07; Primary Completion 2011-01 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The changes of cycloplegic refractive errors | every 6 months for 2 years
  Refractive error was measured using Shin-Nippon NVision-K 5001 autorefractor The changes of cycloplegic objective refractive errors between the treatment and the control were compared.

SECONDARY OUTCOMES:
The changes of axial length | every 6 months for 2 years
  Axial length was measured after cycloplegia using IOL Master

CONTACTS AND LOCATIONS:
Overall Officials: Carly SY Lam, PhD, Principal Investigator — School of Optometry, The Hong Kong PolyU
Locations (1):
- Optometry Clinic, School of Optometry, The Hong Kong PolyU, Hong Kong, China

REFERENCES:
- [Result] Lam CS, Tang WC, Tse DY, Tang YY, To CH. Defocus Incorporated Soft Contact (DISC) lens slows myopia progression in Hong Kong Chinese schoolchildren: a 2-year randomised clinical trial. Br J Ophthalmol. 2014 Jan;98(1):40-5. doi: 10.1136/bjophthalmol-2013-303914. Epub 2013 Oct 29. PMID 24169657
- [Derived] Lawrenson JG, Shah R, Huntjens B, Downie LE, Virgili G, Dhakal R, Verkicharla PK, Li D, Mavi S, Kernohan A, Li T, Walline JJ. Interventions for myopia control in children: a living systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 16;2(2):CD014758. doi: 10.1002/14651858.CD014758.pub2. PMID 36809645